CLINICAL TRIAL: NCT05384899
Title: Central Hub for Kidney Precision Medicine
Brief Title: Kidney Precision Medicine Project (KPMP) - COVID-19 Protocol
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); Icahn School of Medicine at Mount Sinai (Other); Broad Institute of MIT and Harvard (Other); Indiana University (Other); Johns Hopkins University (Other); Joslin Diabetes Center (Other); Pacific Northwest National Laboratory (U.S. Federal Agency); Princeton University (Other); Stanford University (Other); Ohio State University (Other); University of California, San Diego (Other); University of California, San Francisco (Other); The University of Texas Health Science Center at San Antonio (Other); University of Texas (Other); Washington University School of Medicine (Other); Yale University (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Himmelfarb, Professor, School of Medicine, University of Washington
Other Study IDs: SITE00000750 (COV001); 5U2CDK114886 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Failure; Acute Kidney Insufficiency; Acute Renal Failure; Acute Renal Injury; Acute Renal Insufficiency; Kidney Failure, Acute; Kidney Insufficiency, Acute; Renal Failure, Acute; Renal Insufficiency, Acute; Covid19; Sars-CoV-2 Infection
MeSH Terms: conditions — Acute Kidney Injury; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In-hospital blood collection and in-hospital urine collection will be obtained. Collection of remnant kidney (renal) tissue from clinically indicated kidney biopsies in the setting of COVID-19 disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Patients: The focus will be on patients with AKI in the setting of COVID-19 disease.

SUMMARY:
Since its inception, KPMP has developed sophisticated protocols for collection and analysis of human kidney tissue, and for collection of biofluids. Members of the consortium have wide-ranging expertise in conducting clinical studies, processing kidney tissue, advanced structural and molecular analysis and complex bioinformatics analysis, which will be used to leverage effectively as a group to better understand kidney disease.

This joint protocol aims to synergize the COVID-19 study efforts of KPMP academic research centers, to collectively study COVID-19, including its renal presentation using kidney tissue and/or biofluids from patients suffering from COVID-19. This will increase the breadth and depth of data available to the public to expedite discoveries, identify therapeutics, and improve outcomes for patients with COVID-19. It will additionally bring the expertise of KPMP investigators to bear against this pandemic.

DETAILED DESCRIPTION:
The COVID-19 pandemic has drastically altered life globally and killed thousands since its emergence in December of 2019. Unfortunately, the global toll will only continue to increase. Sars-CoV-2, the virus responsible for COVID-19, may directly infect kidney cells, with currently known clinical manifestations of Acute Kidney Injury or nephrotic range proteinuria. Individuals with chronic kidney disease (CKD), diabetes and hypertension are at increased risk of severe COVID-19 infections.

Despite significant effort from industry and academia, development of pharmacologic therapies for AKI and CKD has been hampered by:

Non-predictive animal models The inability to identify and prioritize human targets The limited availability of human kidney biopsy tissue A poor understanding of AKI and CKD heterogeneity Historically, AKI and CKD have been described as single, uniform diseases. However, growing consensus suggests that different disease pathways lead to different subgroups of AKI and CKD (AKIs and CKDs).

Access to human kidney biopsy tissue is a critical first step to define disease heterogeneity and determine the precise molecular pathways that will facilitate identification of specific drug targets and ultimately enable individualized care for people with AKI and CKD.

A number of research centers across the United States are collaborating to bring state-of-the-art technologies together to:

Ethically obtain and evaluate kidney biopsies from participants with AKI or CKD Define disease subgroups Create a kidney tissue atlas Identify critical cells, pathways, and targets for novel therapies

The KPMP is made up of three distinct, but highly interactive, activity groups:

Recruitment Sites: The recruitment sites (RS) are responsible for recruiting participants with AKI or CKD into the longitudinal study and performing the kidney biopsy.

Tissue Interrogation Sites: The tissue interrogation sites (TIS) are responsible for developing and using innovative technologies to analyze the biopsy tissue.

Central Hub: The central hub is responsible for aggregating, analyzing, and visualizing the generated data and providing scientific, infrastructure, and administrative support for the KPMP consortium.

Since its inception, KPMP has developed sophisticated protocols for collection and analysis of human kidney tissue, and for collection of biofluids. Members of the consortium have wide-ranging expertise in conducting clinical studies, processing kidney tissue, advanced structural and molecular analysis and complex bioinformatics analysis, which will be used to to leverage effectively as a group to better understand kidney disease.

This joint protocol aims to synergize the COVID-19 study efforts of KPMP academic research centers, to collectively study COVID-19, including its renal presentation using kidney tissue and/or biofluids from patients suffering from COVID-19. This will increase the breadth and depth of data available to the public to expedite discoveries, identify therapeutics, and improve outcomes for patients with COVID-19. It will additionally bring the expertise of KPMP investigators to bear against this pandemic.

ELIGIBILITY:
Patients 18 years of age or older admitted to participating hospitals with a positive COVID-19 test result or Persons Under Investigation with suspected COVID-19 infection AND with AKI or at high risk of AKI in the setting of COVID-19 infection, as defined by any ONE of the following:

* pre-existing chronic kidney disease as defined by eGFR less than 60 ml/min/1.73 m2
* history of diabetes mellitus established by at least one of the following criteria:

  * Hemoglobin A1C greater than or equal to 6.5%, confirmed with a repeat test within the past year
  * Fasting blood sugar greater than or equal to 126 mg/dL, confirmed with a repeat test within the past year
  * Use of glucose-lowering therapy (insulin or oral or other subcutaneous agents)
  * International Classification of Diseases (ICD) 9/10 diagnostic code for diabetes
* requiring use of vasopressors
* requiring use of mechanical ventilation

AKI is defined by temporal changes in serum creatinine meeting KDIGO Stage 1 criteria or greater (0.3 rise in serum creatinine over baseline value). If a baseline serum creatinine is not available, the patient can be enrolled with an estimated Baseline serum creatinine (see KPMP COVID-19 Manual of Procedures table 1)

Exclusion Criteria:

Any potential participant meeting any one of the general or safety exclusion criteria will not be eligible for enrollment in the KPMP COVID-19 Substudy. Exclusion criteria include non-transient conditions that would not allow for enrollment in the main KPMP study.

Determined at time of Eligibility Assessment prior to consent:

* Non-English or Spanish language
* Less than 18 years of age
* Severe allergy to iodinated contrast
* Transplant recipient (kidney or non-kidney, including solid organ and bone marrow transplantation)
* Additional vulnerable individuals (incarcerated, institutionalized, or otherwise unable to participate in the study)
* Inability to provide informed consent or obtain surrogate consent from a legally authorized representative (LAR)
* Unwilling to receive blood transfusion (if needed)
* Baseline eGFR less than 15 ml/min/m2

If known at the time of enrollment, or determined by kidney ultrasound before the biopsy procedure (may be the same day as the biopsy procedure)

* Kidney size less than 8 cm (percutaneous biopsies only)
* Solitary or single functioning kidney
* Evidence of urinary tract obstruction or hydronephrosis
* Multiple bilateral kidney cysts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The KPMP will focus on COVID-19 positive in-hospital populations that account for large proportions of the public health burden of acute and chronic kidney diseases as evidenced by research and federal data.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Observational: Biorepository of Blood and Urine Specimens | Date of hospital admission through day 28 or hospital discharge [whichever is sooner]. Three month follow-up visit.
  Establish a biorepository of blood and urine specimens from patients with AKI in the setting of COVID-19 disease. For COVID-19 positive patients, in-hospital blood and in-hospital urine are collected within 24 hours of hospital admission. At a follow up visit 3 months after hospital admission, participants will be asked to participate in further bio-specimen collection and/or consent to participate in the main KPMP protocol.
Observational: Biopsy-Related Outcomes | During hospital visit or through study completion if participant wants to enroll into KPMP (up to 10 years, depending on enrollment date of participant)
  For patients who are scheduled for a clinically indicated kidney biopsy in the setting of COVID-19 disease, a segment of remnant tissue may be obtained. We will access the participant's pathology report and store images from their kidney biopsy in the KPMP Digital Pathology Repository. If there is no residual tissue available for analysis, the images will be stored in the KPMP Digital Pathology Repository.
Observational: Phenotypic Clinical Information | Date of hospital admission through day 28 or hospital discharge [whichever is sooner]
  Collection of basic contact information, clinical phenotypic inpatient data relevant to kidney complication of COVID-19 infection, demographics, and linkage to external databases (NDI, USRDS, etc).
Observational: Longitudinal Follow-Up for KPMP Protocol | Through study completion (up to 10 years, depending on enrollment date of participant)
  At a follow-up visit 3 months after hospital admission, participants will be asked to participate in further biospecimen collection and/or consent to participate in the main KPMP protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Texas at Southwestern, Dallas, Texas